CLINICAL TRIAL: NCT06179017
Title: Endovascular Treatment for Mild Stroke With Acute Anterior Circulation Large Vessel Occlusion：a Multicenter Randomized Controlled Trail
Brief Title: Endovascular Treatment for Mild Stroke With Acute Anterior Circulation Large Vessel Occlusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhangzhou Municipal Hospital (Other)
Collaborators: Changhai Hospital (Other); The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Principal Investigator, Wen-huo Chen, Clinical Professor, Zhangzhou Municipal Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MILD-MT
Record Dates: First submitted 2023-12-02; First posted 2023-12-21 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Endovascular Treatment
Keywords: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Intervention group: Endovascular treatment Control group:Best medical treatment
Who Masked: Outcomes Assessor
Masking Description: Endpoint-blined
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group:Endovascular treatment (Experimental): Interventionist choose the optimal EVT strategy and device based on the patient's condition and local guidelines. This may include, but not limited to, stent-retriever thrombectomy, aspiration thrombectomy, intra-arterial thrombolysis, balloon angioplasty, stent implantation and so on. The EVT regimen and relevant time points will be accurately recorded. The patient will receive the best medical treatment according to the local guidelines.
  Interventions: Other: Experimental group:Intervention Group
- Control group: Best medical treatment (Placebo Comparator): Patients will receive the best medical treatment according to local guidelines, including antiplatelet agents, anticoagulants, thrombolysis, etc., but not any EVT. In the control arm, rescue EVT is allowed in patients with disease progression leading to an increase in NIHSS≥4 and excluding the impact of non-stroke factors, and the onset-to-treatment time is within 24 hours.This may include, but not limited to, stent-retriever thrombectomy, aspiration thrombectomy, intra-arterial thrombolysis, balloon angioplasty, stent implantation and so on.
  Interventions: Other: Control group:best medical treatment

INTERVENTIONS:
Other: Experimental group:Intervention Group — Intervention Group:Interventionist choose the optimal endovascular treatment (EVT) strategy and device based on the patient's condition and local guidelines. The patient will receive the best medical treatment according to the local guidelines.
  Arms: Intervention Group:Endovascular treatment
Other: Control group:best medical treatment — Best medical treatment:Patients will receive the best medical treatment according to local guidelines, including antiplatelet agents, anticoagulants, thrombolysis, etc., but not any EVT. In the control arm, rescue EVT is allowed in patients with disease progression leading to an increase in NIHSS≥4 and excluding the impact of non-stroke factors, and the onset-to-treatment time is within 24 hours.
  Arms: Control group: Best medical treatment

SUMMARY:
Exploring the Efficacy and Safety of Emergent Endovascular Treatment in Patients with Mild Ischemic Stroke Caused by Acute Anterior Circulation Large Vessel Occlusion based on Perfusion Imaging Screening

DETAILED DESCRIPTION:
This study aims to select suitable patients with mild AIS caused by anterior circulation LVO with mismatch volume of the ischemic penumbra based on screen of cerebral perfusion imaging. It is a prospective, multicenter, endpoint-blinded, randomized controlled trial design, and aim to explore the efficacy and safety of EVT for mild AIS patients with anterior circulation large vessel occlusion within 24 hours of onset.

ELIGIBILITY:
Inclusion Criteria Inclusion Criteria

1. Age 18-80 years old;
2. Symptoms onset or last known well to randomization is within 24 hours.
3. Clinical diagnosis of acute ischemic stroke due to anterior circulation intracranial large vessel occlusion (LVO) (including intracranial internal carotid artery [ICA], middle cerebral artery [MCA] M1 segment, MCA M2 segment, with or without ipsilateral extracranial ICA occlusion) confirmed on Computerized tomography angiography (CTA) or Magnetic resonance imaging angiography (MRA) ;
4. Baseline NIHSS score <6 before randomization (including cases with NIHSS ≥6 at onset but improves before randomization);
5. ASPECTS score ≥6 based on Non-contrast CT (NCCT) before randomization, and computerized tomography perfusion (CTP) or magnetic resonance imaging perfusion (MRP) imaging presented infarct core volume (relative cerebral blood flow (rCBF) <30%/DWI-ADC<620) ≤50ml, and mismatch volume (Tmax>6 seconds volume - rCBF <30% /DWI-ADC<620) ≥50mL;
6. The patient or their legal representatives voluntarilysigned the informed consent form.

Clinical Exclusion Criteria

1. Premorbid Rankin Scale (mRS) score ≥ 1;
2. Known allergy to iodine, heparin, anaesthesia, or other definite contraindication to receiving endovascular treatment (EVT) procedure;
3. Patient has severe or fatal co-morbidities that could interfere with outcome assessments and follow-up (such as malignant tumor, severe heart failure, or renal failure, or life expectancy less than 6 months);
4. Poorly controlled hypertension (systolic blood pressure >220 mmHg or diastolic blood pressure >120 mmHg);
5. Baseline blood glucose <50mg/dL (2.78 mmol/L) or >400mg/dL (22.20 mmol/L);
6. Known bleeding tendencies, including but not limited to platelet count <100×109/L; received heparin treatment within 48 hours with an activated partial thromboplastin time (APTT) ≥35s; recent oral anticoagulant therapy with international normalized ratio (INR) >3; Note: Patients without a history of coagulation abnormalities or without suspicion of coagulation abnormalities do not need to wait for laboratory test results before enrollment;
7. Seizures at stroke onset or during the course, hard to accurately judge the baseline NIHSS score;
8. Female who is known to be pregnant, lactation, or tested positive for pregnancy at time of admission;
9. Currently participating in another investigational drug study or medical device treatments that may interfere with the results of this study;
10. Other conditions deemed unsuitable for participation, in the opinion of the investigator, or that may pose significant risks to the patient if participating the study.

Imaging Exclusion Criteria:

1. Evidence of intracranial hemorrhage on CT/MRI, including cerebral parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, and subdural/extradural hemorrhage;
2. Significant midline displacement, hernia of brain, or ventricular mass effect with midline displacement confirmed on CT/MRI;
3. Anticipated impossibility to complete endovascular treatment, such as vascular tortuosity, severe vascular wall calcification, etc.;
4. Aortic dissection;
5. Multiple intracranial large vessel occlusions confirmed by CTA or MRA, unable to clearly identify the symptomatic vessel, such as bilateral MCA occlusions or occlusions involving both the MCA and basilar artery;
6. Suspected or confirmed occluded artery is non-acute occlusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
the rate of excellent outcome at () days | 90±7 days and 365±30 days
  mRS score 0-1

SECONDARY OUTCOMES:
mRS shift | 90±7 days and 365±30 days
  distribution of mRS scores
proportion of subjects with good neurological function prognosis | 90±7 days and 365±30 days
  mRS score 0-2

OTHER OUTCOMES:
the rate of symptomatic intracranial hemorrhage | within 48 hours
  according to the Heidelberg criteria
rate of early neurological deterioration | within 7 days
  an increase in NIHSS≥4 or an increase of ≥2 in any individual item
mortality | 90±7 days and 365±30 days
  death

CONTACTS AND LOCATIONS:
Overall Officials: Wenhuo Chen, MD, Study Director — Zhangzhou Municipal Hospital, Zhangzhou Affiliated Hospital of Fujian Medical University
Locations (1):
- Zhangzhou Municipal Hospital, Zhangzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarraj A, Albers GW, Blasco J, Arenillas JF, Ribo M, Hassan AE, de la Ossa NP, Wu TY, Cardona Portela P, Abraham MG, Chen M, Maali L, Kleinig TJ, Cordato D, Wallace AN, Schaafsma JD, Sangha N, Gibson DP, Blackburn SL, De Lera Alfonso M, Pujara D, Shaker F, McCullough-Hicks ME, Moreno Negrete JL, Renu A, Beharry J, Cappelen-Smith C, Rodriguez-Esparragoza L, Olive-Gadea M, Requena M, Almaghrabi T, Mendes Pereira V, Sitton C, Martin-Schild S, Song S, Ma H, Churilov L, Mitchell PJ, Parsons MW, Furlan A, Grotta JC, Donnan GA, Davis SM, Campbell BCV; PERFECT-MILD Collaborators. Thrombectomy versus Medical Management in Mild Strokes due to Large Vessel Occlusion: Exploratory Analysis from the EXTEND-IA Trials and a Pooled International Cohort. Ann Neurol. 2022 Sep;92(3):364-378. doi: 10.1002/ana.26418. Epub 2022 Jul 25. PMID 35599458